CLINICAL TRIAL: NCT00316368
Title: A Study to Determine the Effect of Bi-Ventricular Pacing on Cardiac Hemodynamics After Coronary Artery Bypass Graft
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: 05-318
Record Dates: First submitted 2006-04-18; First posted 2006-04-20 (Estimated); Last update posted 2009-12-23 (Estimated); Status verified 2009-12

CONDITIONS: Coronary Disease
Keywords: Bi-Ventricular pacing post coronary artery bypass graft; coronary artery bypass graft
MeSH Terms: conditions — Coronary Disease

INTERVENTIONS:
Device: Ethicon TPW32 60 cm (pacing wires x 2)

SUMMARY:
The purpose of this study is to determine, using echocardiography, whether bi-ventricular pacing improves the contractile force by resynchronizing both ventricles, thereby improving and/or correcting the paradoxical septal movement.

Primary Hypothesis:

* Bi-ventricular pacing post cardiac surgery will result in at least a 10% increase in cardiac index (CI) as compared with standard atrio-right ventricular pacing.

Secondary Hypothesis:

* Bi-ventricular pacing post cardiac surgery will result in at least a 10% increase in cardiac index (CI) as compared with atrio-left ventricular pacing and right atrium pacing.

DETAILED DESCRIPTION:
Clinical trials done to date have focused on the efficacy of biventricular pacing (BVP) in the treatment of patients with congestive heart failure, Intraventricular conduction delay, dilated cardiomyopathies, and post cardiac surgery. However, studies done in post cardiac surgery patients are limited by their small sample size (4-22 patients with overall of 51 patients), non-randomized pacing protocol and by their inability to determine a definitive mechanism for the improved hemodynamics observed with BVP. Therefore, we propose to complete a pilot study aimed at determining both the magnitude of the hemodynamic benefit associated with BVP, if any. In addition, we will investigate changes in intra-ventricular septal motion as a possible mechanism for the previously observed changes in cardiac hemodynamics.

ELIGIBILITY:
Inclusion Criteria:

* All elective/emergent patients requiring isolated coronary artery bypass graft (CABG) at St. Michael's Hospital.

Exclusion Criteria:

* Patient's age < 18 years.
* Known atrial fibrillation.
* Sinus tachycardia > 100 beats per minute (bpm).
* Post-operative CI < 2.
* High inotrope dosage post-operation:

  * Dopamine (Intropin) if > 10 µg/kg/min.
  * Dobutamine (Dobutrex) if > 10 µg/kg/min.
  * Norepinephrine (Levophed) if > 0.1 µg/kg/min.
  * Epinephrine if > 0.1 µg/kg/min.
* Need for intraaortic balloon pump (IABP).
* Unable or unwilling to give informed consent.
* Already participating in another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-10; Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Cardiac index

SECONDARY OUTCOMES:
Intraventricular motion

CONTACTS AND LOCATIONS:
Overall Officials: David Latter, MD, Principal Investigator — University of Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada